CLINICAL TRIAL: NCT04788862
Title: Open Label Trial to Establish a Blood-stage Controlled Human Malaria Infection Model and Determine Its Safety in Healthy Tanzanian Adults With Varying Prior Exposure to P. Falciparum
Brief Title: A Study of Blood-stage Controlled Human Plasmodium Falciparum Malaria Infection in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Ifakara Health Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VAC083
Record Dates: First submitted 2021-02-25; First posted 2021-03-09 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Malaria; Plasmodium Falciparum
Keywords: Malaria Challenge; Controlled Human Malaria Challenge
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: High prior P. falciparum exposure (Experimental): 6 participants with high previous malaria exposure will be infected via IV administration of Plasmodium falciparum-infected human erythrocytes (planned dose of 1000 iRBCs) of the chloroquine-susceptible 3D7 strain.
  Interventions: Biological: P. falciparum infected erythrocytes
- Group 2: Low prior P. falciparum exposure (Experimental): 6 participants with no or low previous malaria exposure will be infected via IV administration of Plasmodium falciparum-infected human erythrocytes (planned dose of 1000 iRBCs) of the chloroquine-susceptible 3D7 strain.
  Interventions: Biological: P. falciparum infected erythrocytes

INTERVENTIONS:
Biological: P. falciparum infected erythrocytes — Chloroquine sensitive P. falciparum 3D7-infected red blood cells, thawed and prepared under strict aseptic conditions, will be used as a challenge agent.

SUMMARY:
This will be a single-centre, open label trial to determine the safety and feasibility of CHMI model using Plasmodium falciparum-infected cryopreserved erythrocytes administered to healthy Tanzanian adults with varying prior exposure to P. falciparum.

DETAILED DESCRIPTION:
This study will be a single-centre controlled human malaria infection study using adults with varying degrees of prior exposure to P. falciparum. The study will take place at Bagamoyo Clinical Trail Facility of the Ifakara Health Institute, located in Bagamoyo town (about 60 km north of Dar es Salaam).

Twelve healthy male adults aged 18 to 35 years will be recruited into two cohorts of high and low previous exposure consisting of 6 volunteers each as determined by anti-schizont antibody levels. Up to 5 back-up volunteers will be also be recruited and may take the place of another volunteer should they withdraw or become ineligible prior to challenge.

Participants will be infected via IV administration of Plasmodium falciparum-infected human erythrocytes of the chloroquine-susceptible 3D7 strain. Participants will then be closely monitored in a clinical trial facility for a maximum of 31 (28 days plus 3 days of treatment with anti-malarial drugs) days while undergoing frequent clinical and laboratory assessment. Volunteers who do not reach malaria treatment criteria as per protocol at day 28 (C+28) will be treated presumptively with antimalarial medications (ALU + a single low dose primaquine) under direct observation and will be discharged upon completion of treatment and on discretion of the study clinician.

Identifying data will not be included on any trial documentation (other than signed consent) and participants will be referred to by the trial study ID number. The study will be funded primarily by EDCTP grant supporting the evaluation of Multi-Stage Malaria Vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer being adult male aged ≥ 18 and ≤ 35 years, and in good health.
2. Volunteer a resident in Bagamoyo town or rural areas of Bagamoyo district for the past 6 months
3. Able and willing to complete the informed consent process conducted in English
4. Volunteer has adequate understanding of the procedures of the study and is able and willing (in the investigator's opinion) to comply with all study requirements.
5. Volunteer is willing to complete an informed consent questionnaire and is able to answer all questions correctly in a maximum of two attempts.
6. Volunteer is able to communicate well with the investigator and is willing to be monitored in an inpatient setting for 28 days after challenge with infected erythrocytes.
7. The volunteer agrees to refrain from blood donation throughout the study period.
8. Volunteer agrees to refrain from intensive physical exercise (disproportionate to the volunteer's usual daily activity or exercise routine) during the malaria challenge period.
9. Volunteer has signed written informed consent to participate in the trial.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, gastrointestinal, renal, hepatic, neurological, dermatological (e.g. psoriasis, contact dermatitis etc.), allergy, endocrine, malignant, haematological, infectious, immunodeficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results.
2. A heightened risk of cardiovascular disease, as determined by: an estimated ten-year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); history, or evidence at screening, of clinically significant arrhythmia, prolonged QT-interval or other clinically relevant ECG abnormalities; or a positive family history of cardiac events in 1st or 2nd degree relatives <50 years old.
3. Body mass index (BMI) of <18 or >30 Kg/m2
4. A medical history of functional asplenia.
5. History of epilepsy in the period of five years prior to study onset, even if no longer on medication.
6. Confirmed parasite positive by PCR a day before challenge i.e., at C-1.
7. Screening tests positive for Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV)
8. Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral antihistamines exempted) or expected use of such during the study period
9. Any recent or current systemic therapy with an antibiotic or drug with potential antimalarial activity (chloroquine, doxycycline, tetracycline, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, erythromycin, hydroxychloroquine, etc.) (allowable time frame for use at the Investigator's discretion).
10. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.
11. Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.
12. History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
13. Previous participation in any malaria investigational product study (allowable time frame for use at the Investigator's discretion)
14. Known hypersensitivity to or contra-indications (including co-medication) for use of chloroquine, artemether-lumefantrine, Primaquine or history of severe (allergic) reactions to blood transfusion.
15. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
16. Being an employee or relative of an employee of Ifakara Health Institute.
17. Any other condition or situation that would, in the opinion of the investigator, place the volunteer at an unacceptable risk of injury or render the volunteer unable to meet the requirements of the protocol.

Exclusion criteria on day of challenge:

1. Acute disease, defined as moderate or severe illness with or without fever
2. 2. Current COVID-19 infection, defined as ongoing symptoms with positive COVID-19 PCR or rapid antigen test taken during current illness or positive COVID-19 PCR or rapid antigen test within preceding 7 days without symptoms.
3. History of close contact with COVID-19 confirmed case within preceding 14 days

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events to assess the safety of controlled blood-stage P. falciparum | 98 days
  Frequency and severity of clinical and laboratory Adverse Events and Serious Adverse Events
Development of parasitaemia to assess the feasibility of controlled blood-stage P. falciparum | 28 days
  Proportion of participants who develop detectable parasitaemia post-CHMI as measured by qPCR
Development of parasitaemia to assess the feasibility of controlled blood-stage P. falciparum | 28 days
  Proportion of participants who develop sustained parasitaemia detectable by qPCR that is then spontaneously cleared
Parasite multiplication rates to assess the feasibility of controlled blood-stage P. falciparum | 28 days
  Determine parasite multiplication rates as calculated by fitting established models to quantitative PCR data, as routinely done in the published studies (Payne et al., JID 2016; Minassian et al., submitted)

SECONDARY OUTCOMES:
Cellular and Humoral Immune responses level at C-1, C+7, C+14, C+21, C+28, C+56, C+98 and diagnosis | 98 days
  P. falciparum specific immunogenicity following P. falciparum blood-stage infection, as assessed by antibody, B cell and T cell responses. Determined by ELISA (concentration of antibodies)
Cellular and Humoral Immune responses level at C-1, C+7, C+14, C+21, C+28, C+56, C+98 and diagnosis | 98 days
  P. falciparum specific immunogenicity following P. falciparum blood-stage infection, as assessed by antibody, B cell and T cell responses. Determined by ELISpot (spots per 10^x PBMCs)
Cellular and Humoral Immune responses level at C-1, C+7, C+14, C+21, C+28, C+56, C+98 and diagnosis | 98 days
  P. falciparum specific immunogenicity following P. falciparum blood-stage infection, as assessed by antibody, B cell and T cell responses. Determined by flow cytometry (% of immune cell sub-population)
To determine the effect of pre-exposure to malaria on parasite multiplication rates following controlled blood-stage P. falciparum infection. | 28 days
  Comparison of PMRs between participants with low and high prior exposure to P. falciparum.
To determine if malaria infection following inoculation of P. falciparum is caused by the inoculum parasite strain and not wild-type strains | 28 days
  Determine whole genome sequences (via whole genome analysis) following controlled blood-stage P. falciparum infection to confirm malaria infection is with inoculum strain and not wild-type parasite

CONTACTS AND LOCATIONS:
Overall Officials: Angela Minassian, Dr, Principal Investigator — University of Oxford
Locations (1):
- Ifakara Health Institute, Bagamoyo, Tanzania